CLINICAL TRIAL: NCT00002002
Title: A Randomized, Double-Blind, Placebo Controlled Study of l-Leucovorin in Combination With Trimethoprim / Sulfamethoxazole in the Therapy of Pneumocystis Carinii Pneumonia in Patients With the Acquired Immunodeficiency Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lederle Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 056A; 76-9
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-07

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Trimethoprim; Sulfamethoxazole; Leucovorin

INTERVENTIONS:
Drug: Trimethoprim
Drug: Sulfamethoxazole
Drug: Leucovorin calcium

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of l-leucovorin in preventing toxicity from high dose trimethoprim / sulfamethoxazole (TMP / SMX) used as a therapy for Pneumocystis carinii pneumonia (PCP) in patients with AIDS.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Diagnosis of PCP.
* Fit the CDC definition of AIDS.
* Be receiving intravenous or oral trimethoprim / sulfamethoxazole (Bactrim, Septra) in doses of = or > 15mg/kg/day of the trimethoprim component.
* Be receiving = or < 48 hours of trimethoprim / sulfamethoxazole (TMP / SMX) prior to randomization.
* Must sign informed consent in accordance with FDA guidelines.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Cannot take oral medications.
* Require continued administration of anticonvulsant agents such as phenytoin, phenobarbital or primidone.

Concurrent Medication:

Excluded:

* Continued administration of anticonvulsant agents such as phenytoin, phenobarbital or primidone.

Patients with the following are excluded:

* Cannot take oral medications.
* Require continued administration of anticonvulsant agents such as phenytoin, phenobarbital or primidone.

Prior Medication:

Excluded:

* > 48 hours of trimethoprim / sulfamethoxazole prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Gen Hosp, San Francisco, California, United States

REFERENCES:
- [Background] Safrin S, Lee BL, Sande MA. Adjunctive folinic acid with trimethoprim-sulfamethoxazole for Pneumocystis carinii pneumonia in AIDS patients is associated with an increased risk of therapeutic failure and death. J Infect Dis. 1994 Oct;170(4):912-7. doi: 10.1093/infdis/170.4.912. PMID 7930736